CLINICAL TRIAL: NCT06800729
Title: A Single Center, Single Dose, Randomized, Placebo-controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Orally Administered TIX100 in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate Safety, Tolerability and Pharmacokinetics of TIX100 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TIXiMED, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIX100-01
Record Dates: First submitted 2025-01-23; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: TIX100; TIXiMED; inhibitor of thioredoxin-interacting protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- TIX100 20 mg (Active Comparator)
  Interventions: Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein
- TIX100 60 mg (Active Comparator)
  Interventions: Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein
- TIX100 100 mg (Active Comparator)
  Interventions: Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein
- TIX100 160 mg (Active Comparator)
  Interventions: Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein
- TIX100 200 mg (Active Comparator)
  Interventions: Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TIX100, an orally available inhibitor of thioredoxin-interacting protein — TIX100, an orally available inhibitor of thioredoxin-interacting protein
  Arms: TIX100 100 mg; TIX100 160 mg; TIX100 20 mg; TIX100 200 mg; TIX100 60 mg
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
A Single Center, Single Dose, Randomized, Placebo-controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Orally Administered TIX100 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 years, both genders.
2. Healthy as determined by a physician, based on history, medical examination, vital signs, laboratory tests, cardiac monitoring and respiratory function. History must comply with the following:

   1. Absence of clinically significant illness or surgery within the preceding 12 weeks.
   2. Absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and/or metabolic disease.
3. Male subjects with female partners of childbearing potential must agree to utilize condoms for the duration of the study.
4. Female subjects of child-bearing potential with negative urine pregnancy tests and who agree to use double-barrier contraception during the study. The primary contraception may be either hormonal implant or hormonal or non-hormonal intrauterine device, and the secondary (barrier) method of contraception with condom and/or with spermicide.
5. Female subjects of non-child-bearing potential (i.e. tubal ligation, hysterectomy, or postmenopausal).
6. Body mass index (BMI) 18.5 - 29.9 kg/m2
7. HbA1c <6.0%

Exclusion Criteria:

1. History of excessive alcohol use (defined as >21 drinks per week for males and >14 drinks per week for females), recreational drug use or drugs of abuse within the past three months, or failure on urinary drug screen.
2. Pregnant or breastfeeding within six months of screening assessment.
3. Substantial changes in eating habits or exercise routine within the preceding three months.
4. Evidence of eating disorders.
5. >5% weight change in the past three months.
6. Bariatric surgery within the past five years.
7. Significant renal impairment (eGFR <60 mg/mL/1.73m2).
8. Liver function tests (i.e., ALT, AST, alkaline phosphatase) greater than twice the upper limit of normal upon repeated measurements.
9. Diseases interfering with metabolism and/or ingestive behavior (e.g., myxedema, Cushing's disease, schizophrenia, major psychoses, unmanaged depression).
10. Use of drugs approved for the treatment of obesity.
11. Any clinically significant abnormality following the Investigator's review of the physical examination and clinical laboratory tests.
12. A baseline prolongation of QT/QTc interval after repeated measurements of >450 ms; a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of LQTS.
13. Participation in an investigational drug trial within three months prior to dosing in the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 7
Number of participants with laboratory analyte results above upper limit of normal. | Day 7
Number of participants with vital sign results considered clinically significant by the investigator | Day 7
Number of participants with ECG results considered clinically significant by the investigator | Day 7
Number of participants with physical examination findings considered clinically significant by the investigator | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No
Phase 1 healthy volunteer study